CLINICAL TRIAL: NCT04865302
Title: Cerebral Oxygenation in Preterm Neonates with Respiratory Support During Skin-to-skin Care on the First Day After Birth - a Prospective Observational Pilot Study
Brief Title: Cerebral Oxygenation in Preterm Neonates with Respiratory Support During Skin-to-skin Care on the First Day After Birth
Acronym: Kangaroo
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Kangaroo
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2023-11

CONDITIONS: Preterm Birth; Ventilator Lung; Newborn
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: SSC — Incubator phase I: After feeding the neonates will be brought in a prone position in the incubator and the NIRS sensor will be applied on the forehead for continuous cStO2 measurements throughout the study period. The neonate will rest in this position for 60 minutes.
  SSC phase: The neonate will be brought on the mother's or father's chest (skin to skin) in a prone position and will stay in this position for 60 minutes.
  Incubator phase II: The neonates will be brought back into the incubator for another 60 minutes in prone position. After 180 minutes the study period is over and the NIRS sensor will be removed.

SUMMARY:
This is a prospective observational pilot study investigating if skin-to-skin care (SSC) has an influence on cerebral oxygenation and perfusion measured with near-infrared spectroscopy (NIRS) compared to incubator care in ventilated preterm neonates on the first day after birth.

DETAILED DESCRIPTION:
Background

Kangaroo mother care (KMC) or skin-to-skin care (SSC) is a routine method of care in preterm neonates in neonatal intensive care units around the world. SSC is mostly defined as the skin-to-skin contact of the infant with the mother's or father's chest, which has been proven to reduce mortality, decrease severe illness, nosocomial infections and the length of hospital stay as well as to improve growth, breastfeeding and mother-child-relationship. During the last years several studies were performed showing that SSC provides comparable neonatal physiological stability compared to routine incubator care.

Near-infrared spectroscopy (NIRS) enables non-invasive, continuous monitoring of oxygenation and perfusion in different tissues. Several studies have shown that SSC has no negative influence on cerebral oxygenation saturation and physiological parameters compared to routine incubator care in preterm infants with respiratory support after the 5th day after birth. Nevertheless, until now there is no information on cerebral oxygenation and physiological parameters during SSC compared to routine incubator care in preterm neonates with respiratory support during the first 24 hours after birth, when transition still takes place and may cause unstable vital signs in neonates. Cerebral hypoxia as well as hyperoxia can cause severe brain damage due to perfusion disturbances, especially in ventilated preterm neonates.

Objectives

Primary aim: To assess, if the burden of cerebral hypoxia (calculated as the area under the curve outside the tissue oxygenation (cStO2) target range of 55% - 76%) in preterm neonates with respiratory support is different during SSC compared to routine incubator care on the first day after birth.

Secondary aims: To assess, if SSC has an influence on cFTOE (cerebral fractional tissue oxygen extraction) and routine monitoring parameters (arterial oxygen saturation [SpO2], heart rate [HR], respiratory rate [RR], mean arterial blood pressure [MABP], temperature) in preterm neonates with respiratory support compared to routine incubator care on the first day after birth.

Methods

Study population: Preterm neonates <37+0 weeks of gestation with respiratory support admitted to the Division of Neonatology, Department of Paediatrics and Adolescent Medicine, Medical University of Graz after vaginal delivery or caesarean section will be eligible for the study.

Procedure: Patients and maternal medical history and main diagnoses, as well as routinely sampled laboratory results, provided therapy and respiratory support will be documented in each neonate.´

Measurements: For NIRS measurements the OxyPrem 1.4. (OxyPrem AG, Zurich, Switzerland) will be used. The NIRS measurements will take place once during the first day after birth before / during / after routine SSC and will last for 180 minutes.

After feeding the neonates will be brought in a prone position in the incubator and the NIRS sensor will be applied on the forehead for continuous cStO2 measurements throughout the study period. The neonate will rest in this position for 60 minutes. Afterwards the neonate will be brought on the mother's or father's chest (skin to skin) in a prone position and will stay in this position for 60 minutes. Finally the neonates will be brought back into the incubator for another 60 minutes in prone position. After 180 minutes the study period is over and the NIRS sensor will be removed.

Furthermore, NIRS will be combined with routine monitoring, such as pulse oxymetry (SpO2, HR), blood pressure measurements and measurements of temperature. Data will be stored in a polygraphic system (alpha-trace digitalMM, B.E.S.T. Medical Systems, Austria) for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Need for respiratory support (endotracheal tube [ETT], nasal continuous positive airway pressure [nCPAP], high-flow nasal cannula [HFNC])
* Decision to conduct full life support
* Written informed consent

Exclusion Criteria:

* No decision to conduct full life support
* No written informed consent
* Severe congenital malformations, severe asphyxia (umbilical cord artery pH <7.00)
* Cerebral malformations, posthaemorrhagic ventricular dilatation, intraventricular haemorrhage grade III, periventricular haemorrhage
* Cardiovascular instability (need for catecholamines)
* No need for respiratory support

Ages: 15 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates <37+0 weeks of gestation admitted to the Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz after vaginal delivery or caesarean section will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
percent minutes of cerebral hypoxia | 60 minutes
  After a 20 minutes washout period the time (percentage of minutes) of cerebral hypoxia (below 54%) will be calculated for intervention period "incubator phase I" over 40 minutes.
percent minutes of cerebral hypoxia | 60 minutes
  After a 20 minutes washout period the time (percentage of minutes) of cerebral hypoxia (below 54%) will be calculated for intervention period "SSC" over 40 minutes.
percent minutes of cerebral hypoxia | 60 minutes
  After a 20 minutes washout period the time (percentage of minutes) of cerebral hypoxia (below 54%) will be calculated for intervention period "incubator phase II" over 40 minutes.

SECONDARY OUTCOMES:
Mean StO2 | 60 minutes
  Mean StO2 values over 40 minutes, calculated for intervention period "incubator phase I", after washout time will be calculated
Mean StO2 | 60 minutes
  Mean StO2 values over 40 minutes, calculated for intervention period "SSC", after washout time will be calculated
Mean StO2 | 60 minutes
  Mean StO2 values over 40 minutes, calculated for intervention period "incubator phase II" after washout time will be calculated
Mean cFTOE | 60 minutes
  Mean cFTOE values over 40 minutes for intervention period "incubator phase I" after washout time will be calculated
Mean cFTOE | 60 minutes
  Mean cFTOE values over 40 minutes for intervention period "SSC" after washout time will be calculated
Mean cFTOE | 60 minutes
  Mean cFTOE values over 40 minutes for intervention period "incubator phase II" after washout time will be calculated
Mean routine monitoring parameters :SpO2 | 60 minutes
  SpO2 for intervention period "incubator phase I"
Mean routine monitoring parameters :SpO2 | 60 minutes
  SpO2 for intervention period "SSC"
Mean routine monitoring parameters :SpO2 | 60 minutes
  SpO2 for intervention period "incubator phase II"
Mean routine monitoring parameters: HR | 60 minutes
  HR for intervention period "incubator phase I"
Mean routine monitoring parameters: HR | 60 minutes
  HR for intervention period "SSC"
Mean routine monitoring parameters: HR | 60 minutes
  HR for intervention period "incubator phase II"
Mean routine monitoring parameters: RR | 60 minutes
  RR for intervention period "incubator phase I"
Mean routine monitoring parameters: RR | 60 minutes
  RR for intervention period "SSC"
Mean routine monitoring parameters: RR | 60 minutes
  RR for intervention period "incubator phase II"
Mean routine monitoring parameters: MABP | 60 minutes
  MABP for intervention period "incubator phase I"
Mean routine monitoring parameters: MABP | 60 minutes
  MABP for intervention period "SSC"
Mean routine monitoring parameters: MABP | 60 minutes
  MABP for intervention period "incubator phase II"
Mean routine monitoring parameters: temperature | 60 minutes
  Temperature for intervention period "incubator phase I"
Mean routine monitoring parameters: temperature | 60 minutes
  Temperature for intervention period "SSC"
Mean routine monitoring parameters: temperature | 60 minutes
  Temperature for intervention period "incubator phase II"

OTHER OUTCOMES:
leukocyte count | first 48 hours
  leukocyte count (per µl) - routinely sampled
C-reactive protein | first 48 hours
  C-reactive protein (mg/l) - routinely sampled
IT-ratio | first 48 hours
  IT-ratio - routinely sampled

CONTACTS AND LOCATIONS:
Overall Officials: Nina Höller, MD, Principal Investigator — Medical University of Graz, Department of Paediatrics and Adolescent Medicine, Devision of Neonatology
Locations (1):
- Department of Pediatrics, Division of Neonatology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No